CLINICAL TRIAL: NCT03818594
Title: Challenges in Achieving Adequate Vitamin D Status in the Adult Population - Part 1
Acronym: VITAD/1
Status: Completed | Type: Observational
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: VIST - Faculty of Applied Sciences (Other); Slovenian Research Agency (Other); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Sponsor
Other Study IDs: VITAD-01-2018 Part 1
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Serum Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Seasonal variations in vitamin D status will be determined on a cohort of Slovenian adults using longitudinal study design, and association between vitamin D status and different Caucasian phototypes, skin colour and melanin index investigated .

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent form (ICF),
* Caucasian race
* Age between 18 and 65 years at the time of the signature of Informed consent form (ICF),
* Willingness to avoid a consumption of any food supplements containing Vitamin D during the study, except the ones prescribed by the study researchers, and to avoid use of solarium or other artificial UVB sources
* Willingness to follow all study procedures

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products in Part 2,
* Pronounced avoidance of sunshine (eg reporting of allergy to the sun)
* Use of food supplements containing Vitamin D or fish oil or omega 3 fatty acids in last three months prior to inclusion,
* Special dietary habits used by a small part of the population (veganism, low-carb hihg-fat diet, caloric restriction diet, note: vegetarians are not excluded)
* Diets prescribed by the medical profession
* Disorders of the kidneys, thyroid, digestive tract, osteoporosis and other bone diseases, skin diseases
* Other diseases and conditions that affect the absorption and synthesis of vitamin D
* Exposure to stronger sunlight in the last three months prior to engaging in a survey (travel to countries with stronger sunshine, use of solarium),
* The consumption of margarine or plant substitutes for milk / milk products several times a day, as these foods are most often enriched with vitamin D,
* Visiting the solarium in the last three months before joining the survey,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Slovenian adult population, men and women, skin phototypes I-IV.
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Difference between vitamin D serum levels in winter and in summer season will be determined | 2 years
  Vitamin D serum level will be measured once in winter (December - January) and once in summer season (August-September) for each individual. The study will be performed over two consecutive years.

SECONDARY OUTCOMES:
Correlation of vitamin D serum levels with Fitzpatrick skin phototype | 2 years
  Fitzpatrick skin phototype will be determined using Fitzpatrick self-evaluation questionnaire in combination with expert assessment in August-September.
Correlation of vitamin D serum levels with skin colour measured in CIE Lab colour space | 2 years
  Skin colour will be measured in CIE Lab colour space on inner and outer side of the upper arm. The measurement will be performed in August-September.
Correlation of vitamin D serum levels with melanin index | 2 years
  Melanin index will be measured on inner and outer side of the upper arm. The measurement will be performed in August-September.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Principal Investigator — Researcher
Locations (1):
- Nutrition Institute, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No